CLINICAL TRIAL: NCT06570083
Title: Mobile-Based Intervention to Promote Physical Activity Among the Elderly With Chronic Diseases
Brief Title: Mobile-Based Intervention to Promote Physical Activity Among the Elderly
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mobile Elderly Exercise
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Mobile Health; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will receive three months of personalized support via WeChat, including tailored exercise recommendations, motivational messages, and educational content.
  Interventions: Behavioral: Mobile Exercise Support; Behavioral: Self-help physical activity booklet
- Control group (Active Comparator): Participants in the control group will receive a self-help booklet designed to promote physical activity among the elderly.
  Interventions: Behavioral: Self-help physical activity booklet

INTERVENTIONS:
Behavioral: Mobile Exercise Support — Participants receive three months of personalized support via WeChat, including tailored exercise recommendations, motivational messages, and educational content.
  Arms: Intervention group
Behavioral: Self-help physical activity booklet — Participants receive a self-help booklet to promote physical activity among the elderly. The booklet will include guidelines for safe and effective exercises, tips for staying motivated, and information on the health benefits of regular physical activity.

SUMMARY:
This study aims to explore the feasibility and preliminary effectiveness of a mobile phone-based intervention among elderly individuals with chronic diseases.

DETAILED DESCRIPTION:
Promoting physical activity among elderly individuals is an increasingly critical public health priority. Regular exercise is essential for maintaining mobility, enhancing mental well-being, and reducing the risk of exacerbating chronic conditions. However, many elderly individuals encounter significant barriers, including physical limitations, lack of motivation, and restricted access to safe environments.

This mobile phone-based intervention seeks to address these challenges by offering accessible support through age-appropriate exercise routines, motivational prompts, and educational content delivered directly to participants' mobile devices. The intervention's primary objective is to reduce sedentary behavior, increase physical activity levels, and ultimately enhance the overall health and well-being of elderly individuals with chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥60 years and diagnosed with at least one chronic disease
2. Owns a smartphone and is proficient in using WeChat
3. Daily sedentary time ≥6 hours

Exclusion Criteria:

1. recent surgeries, injuries, or other conditions that would prevent simple physical activity
2. hearing, vision, or physical disabilities

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Time spent in sedentary behavior | 3 and 6 months follow-up
  The time spent sedentary behavior (min/week) in the last 7 days
Acceptability of the Mobile Phone-Based Intervention | 3 and 6 months follow-up
  Acceptability will be assessed using a series of 4 items from previous studies on mobile physical activity interventions. Participants will rate each statement on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). The statements will cover aspects such as ease of use, personal relevance, clarity of information, and overall satisfaction with the intervention.
Perceived Usefulness of the Mobile Phone-Based Intervention | 3 and 6 months follow-up
  Perceived usefulness will be assessed using 5 items from previous studies on online physical activity interventions. Participants will rate each question on a 5-point Likert scale, ranging from 1 (not at all useful) to 5 (very useful). The questions will explore how useful participants found the intervention in helping them to (1) increase confidence in engaging in regular physical activity, (2) overcome barriers to physical activity, (3) increase support for participating in physical activity, (4) plan for physical activity, and (5) stay motivated to engage in physical activity.

SECONDARY OUTCOMES:
Time spent in zero-time exercise | 3 and 6 months follow-up
  The time spent physical activity while seated and standing (min/week) in the last 7 days
Exercise self-efficacy | 3 and 6 months follow-up
  This outcome measure evaluates participants' confidence in their ability to engage in regular physical activity (self-efficacy). Participants will rate their confidence on a single-item scale ranging from 1 to 10, with higher scores indicating greater self-efficacy.
Anxiety and depression | 3 and 6 months follow-up
  Anxiety and depression levels will be assessed using the Patient Health Questionnaire-4 (PHQ-4), a validated tool comprising two items for anxiety and two items for depression. The PHQ-4 score ranges from 0 to 12, with higher scores indicating greater severity of anxiety and depression symptoms.
Perceived subjective happiness | 3 and 6 months follow-up
  This outcome measure assesses participants' subjective happiness using a Self-Reported Happiness scale. Participants will rate their happiness on a single-item scale ranging from 1 (not at all happy) to 5 (extremely happy), with higher scores indicating greater perceived happiness.
Perceived life satisfaction | 3 and 6 months follow-up
  This outcome measure assesses participants' subjective life satisfaction using a self-reported life satisfaction scale. Participants will rate their life satisfaction on a single-item scale ranging from 1 to 5, with higher scores indicating greater perceived life satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Normal University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No